CLINICAL TRIAL: NCT03209167
Title: Comparing Patient Satisfaction of the Abdomen After DIEAP Procedure and Conventional Abdominoplasty
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kim Alexander Tønseth, Head of division, Oslo University Hospital
Other Study IDs: OsloPlastic
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Donor Site Complication; Satisfaction, Personal; Breast Cancer
Keywords: Breast reconstruction; abdominoplasty; patient satisfaction
MeSH Terms: conditions — Personal Satisfaction; Breast Neoplasms; Patient Satisfaction | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DIEAP group: Patients who had undergone DIEAP flap breast reconstruction
  Interventions: Behavioral: Questionnaire
- AP group: Patients who had undergone conventional abdominoplasty
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Two study-specific questionnaires

SUMMARY:
The purpose of this study was to specifically compare the long term patient satisfaction of the abdomen after DIEAP flap procedure with conventional abdominoplasty.

DETAILED DESCRIPTION:
34 patients reconstructed with a DIEAP flap (DIEAP group) and 30 patients who had undergone a conventional abdominoplasty (AP group) were asked to complete two study-specific questionnaires. One questionnaire covered general and specific aspects concerning abdominal outcomes and morbidity. The other covered general outcomes such as satisfaction with surgery and change of body image, self-confidence, social and intimate relations. In addition, all patients performed an abdominal muscle function test.

ELIGIBILITY:
Inclusion Criteria:

* unilateral DIEAP flap, abdominoplasty

Exclusion Criteria:

* bilateral DIEAP flap, progressive cancer disease

Age Groups: Child, Adult, Older Adult
Enrollment: 44
Dates: Start 2001-01-01 (Actual); Primary Completion 2004-12-31 (Actual); Study Completion 2004-12-31 (Actual)

PRIMARY OUTCOMES:
Comparing patient satisfaction of the abdomen after DIEAP procedure and conventional abdominoplasty | 2001 to 2004.
  The purpose of this study was to specifically compare the long term patient satisfaction of the abdomen after DIEAP flap procedure with conventional abdominoplasty.